CLINICAL TRIAL: NCT07343037
Title: Diagnosis of Lymphohistiocytic Hemophagocytosis in Intensive Care: Relevance of the Hscore and Search for the Best Diagnostic Markers
Brief Title: Diagnosis of Lymphohistiocytic Hemophagocytosis in Intensive Care
Acronym: SAMICU
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9818
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Insufficiency; Cirrhosis, Liver
Keywords: Hepatic Insufficiency; Cirrhosis, Liver; Lymphohistiocytic hemophagocytosis; Hepatocellular insufficiency; Invasive aspergillosis; Azole antifungals; Liver dysfunction.
MeSH Terms: conditions — Hepatic Insufficiency; Liver Cirrhosis; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with hepatocellular insufficiency and/or cirrhosis are at risk of developing invasive fungal infections, particularly in critical care settings.

In international recommendations, voriconazole is positioned as the first-line treatment for invasive aspergillosis. However, this molecule-and the azole class of antifungals-is associated with frequent hepatic toxicity. Available since 2018, isavuconazole appears to be better tolerated in patients without pre-existing liver dysfunction.

The aim of this study is to retrospectively evaluate the validity of the hscore in intensive care and resuscitation patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Patient admitted to the intensive care unit at Hautepierre Hospital, Strasbourg University Hospital, between January 1, 2014, and December 31, 2024
* At least 3 biological signs of HLH:

  * ferritin > 2000 ng/mL
  * triglycerides > 1.5 g/L
  * at least one cytopenia (leukocytes ≤ 5000 G/L, platelets ≤ 110 G/L, hemoglobin ≤ 9.2 g/dL).

Exclusion Criteria:

Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient admitted to the intensive care unit at Hautepierre Hospital, Strasbourg University Hospital, between January 1, 2014, and December 31, 2024
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
hscore | Up to 12 months
  The HScore adds up points assigned to 9 clinical, biological, and histological criteria:
  The higher the total score, the greater the likelihood of HLH:
  Possible total score: 0 to 337:
  HScore: Probability of HLH:
  < 90 points → Very low
  * 130 points → ≈ 10-20% 168 points → high probability of HL

CONTACTS AND LOCATIONS:
Locations (1):
- Médecine intensive - Réanimation - CHU de Strasbourg - France, Strasbourg, France